CLINICAL TRIAL: NCT07101666
Title: Total Neoadjuvant Therapy With Short Course Radiation Therapy in Gastric Cancer
Acronym: TNT-SHORT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-x143
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; SCRT
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SCRT + SOC Neoadjuvant Chemotherapy (Experimental): Patients will be treated with short course radiation therapy (SCRT) followed by 4 months of standard of care (SOC) neoadjuvant chemotherapy. Patients will then undergo gastrectomy (if medically operable) or surveillance (if medically inoperable).
  Interventions: Radiation: Short course radiation therapy; Drug: Standard of care neoadjuvant chemotherapy

INTERVENTIONS:
Radiation: Short course radiation therapy — 25 Gy in 5 fractions
  Other Names: SCRT
Drug: Standard of care neoadjuvant chemotherapy — Recommended options are CAPOX, FOLFOX, or FLOT but other standard of care chemotherapy may be given given at the discretion of the treating medical oncologist after consultation with the study Principal Investigator.

SUMMARY:
Standard treatment for patients with early stage gastric cancer consists of perioperative chemotherapy and surgical resection. If radiation therapy is administered in the adjuvant setting, the radiated area is often large and associated with significant toxicity.

In this study, the investigators propose the addition of short course radiation therapy (SCRT) to chemotherapy in the neoadjuvant setting. The investigators hypothesize that this regimen of Total Neoadjuvant Therapy (TNT) will result in a higher rate of complete response (both pathologic and clinical), with less toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed histologically or cytologically gastric adenocarcinoma. (Siewert III acceptable: the bulk of tumor should be in stomach; gastric tumors with extension to the gastroesophageal junction are permitted.) Patients with T1-4N0-3 are eligible.
* Known T-stage defined by EUS. Must have had CT of the chest/abdomen/pelvis with IV contrast (or PET/CT if unable to receive iodinated contrast).
* Medically eligible to receive SOC chemotherapy.
* At least 18 years of age.
* ECOG performance status ≤ 2.
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Creatinine clearance > 50 mL/min by Cockroft Gault calculation
* The effects of the various chemotherapy agents used in this study on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and one month after completion of the study.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Prior surgery, radiation, or chemotherapy for gastric or esophageal cancer.
* Prior surgery to the esophagus or stomach.
* Siewert I-II GE junction tumor.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to the SOC chemotherapy used in the study.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia that are considered clinically significant as determined by the treating physician.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days of study entry.
* HIV-infected if not on effective anti-retroviral therapy with undetectable viral load for 6 months. Patients with HIV who are receiving effective anti-retroviral therapy and have had an undetectable viral load for at least 6 months are eligible. HIV testing not required in the absence of known history of infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | Through completion of surgery (estimated to be 6 months) for operable patients or through 12 months after end of treatment for inoperable patients (estimated to be 18 months)
  Complete response is defined as pathologic complete response (pCR) in operable patients and durable (1-year) clinical complete response (cCR) in medically inoperable patients.
  * pCR in operable patients is defined as no tumor on gastrectomy specimen.
  * Clinical complete response rate in inoperable patients is defined as having no evidence of disease on EUS and/or EGD and no definite evidence of disease on PET/CT.

SECONDARY OUTCOMES:
Rate of grade 3 or greater adverse events as defined by CTCAE v 5.0 | From day 1 of SCRT through 12 months after surgery/definitive end of treatment (estimated to be 18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Grierson, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - UCLA, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu